CLINICAL TRIAL: NCT01195259
Title: A Meta Analysis of Malignancy Serious Adverse Events in the ADOPT, 49653/048, and RECORD, 49653/231, Studies, Comparing Metformin With Rosiglitazone.
Brief Title: Malignancy Meta Analysis for BRL49653
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114769
Record Dates: First submitted 2010-09-01; First posted 2010-09-06 (Estimated); Last update posted 2013-10-28 (Estimated); Status verified 2013-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: rosiglitazone; ADOPT; metformin; malignancy; RECORD
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Neoplasms | interventions — Metformin; Rosiglitazone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- metformin: Subjects from ADOPT that are included in this meta-analysis were randomly allocated to receive metformin or rosiglitazone. Subjects from RECORD that are included in this meta-analysis were taking one of three sulfonylureas (glibenclamide, gliclazide or glimepiride) and were randomly allocated metformin or rosiglitazone to use as add-on treament to background sulfonylurea.
  Interventions: Drug: allocation of treatment with metformin or rosiglitazone
- rosiglitazone: Subjects from ADOPT that are included in this meta-analysis were randomly allocated to receive metformin or rosiglitazone. Subjects from RECORD that are included in this meta-analysis were taking one of three sulfonylureas (glibenclamide, gliclazide or glimepiride) and were randomly allocated metformin or rosiglitazone to use as add-on treament to background sulfonylurea.
  Interventions: Drug: allocation of treatment with metformin or rosiglitazone

INTERVENTIONS:
Drug: allocation of treatment with metformin or rosiglitazone — Subjects from ADOPT that are included in this meta-analysis were randomly allocated to receive metformin or rosiglitazone. Subjects from RECORD that are included in this meta-analysis were taking one of three sulfonylureas (glibenclamide, gliclazide or glimepiride) and were randomly allocated metformin or rosiglitazone to use as add-on treament to background sulfonylurea.

SUMMARY:
Observational analyses of data from population registeries have suggested that metformin may be associated with a decreased prevalence of malignancy. The ADOPT and RECORD studies both contain groups of subjects randomly allocated to metformin and rosiglitazone. This meta-analysis combines malignancy serious adverse events from ADOPT and RECORD in order to compare their incidence on metformin with that on rosiglitazone.

DETAILED DESCRIPTION:
The objective of this meta-analysis is to compare the incidence of malignancy (excluding non-melanomatous skin cancers) reported as serious adverse events in the ADOPT and RECORD studies between subjects randomly allocated to treatment with metformin with those allocated to rosiglitazone.

ELIGIBILITY:
Subjects from ADOPT that are included in this meta-analysis (those in the metformin or rosiglitazone groups) had the dose of their study medication increased to a maximum of 2g (metformin) or 8mg (rosiglitazone) if their fasting plasma glucose was greater than 140mg/dl.

Subjects from RECORD that are included in this meta-analsyis entered the RECORD study taking one of three sulfonylureas (glibenclamide, gliclazide or glimepiride). They were randomly allocated to metformin or rosiglitazone in a 1:1 ration to use as add-on treatment to the background of sulfonylurea. These subjects had the dose of their study medication increased to a maximum of 2.55g (metformin) or 8mg (rosiglitazone) if their HbA1c was greater than 7.0%.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 5135 subjects with type 2 diabetes mellitus from the intention to treat (ITT) populations of 2 randomised, controlled studies (2576 metformin/2559 rosiglitazone)
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2009-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Time to first occurrence of a serious adverse event of malignancy (excluding non-melanomatous skin cancers) | ADOPT approximately 4 years duration, RECORD approximately 5.5 years duration

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Background] Home PD, Kahn SE, Jones NP, Noronha D, Beck-Nielsen H, Viberti G; ADOPT Study Group; RECORD Steering Committee. Experience of malignancies with oral glucose-lowering drugs in the randomised controlled ADOPT (A Diabetes Outcome Progression Trial) and RECORD (Rosiglitazone Evaluated for Cardiovascular Outcomes and Regulation of Glycaemia in Diabetes) clinical trials. Diabetologia. 2010 Sep;53(9):1838-45. doi: 10.1007/s00125-010-1804-y. Epub 2010 Jun 8. PMID 20532476